CLINICAL TRIAL: NCT03285841
Title: Co-registered Multimodal Optical Imaging for the Early Detection and Management of Cancers of the Vulva and Cervix
Brief Title: OCT-AF Imaging of Pre-cancers of Vulva and Cervix
Status: Terminated | Type: Observational
Why Stopped: No funding
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: BCCR-H17-02004
Record Dates: First submitted 2017-09-12; First posted 2017-09-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Cervical Dysplasia; Vulvar Dysplasia; Precancerous Lesions; Vulvar Cancer; Cervical Cancer
Keywords: cervical cancer; vulvar cancer; optical coherence tomography; autofluorescence imaging
MeSH Terms: conditions — Uterine Cervical Dysplasia; Vulvar Neoplasms; Uterine Cervical Neoplasms | interventions — Multimodal Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cervical Sites: Imaging complete cervix from endocervical canal to transformation zone to ectocervix.
  Interventions: Device: OCT-AFI
- Vulvar sites: Imaging vulvar lesions
  Interventions: Device: OCT-AFI

INTERVENTIONS:
Device: OCT-AFI — Both groups will be imaged with the OCT-AFI device. Imaging will not influence standard of care biospies, treatment and procedures.
  Other Names: Multimodal imaging

SUMMARY:
The multimodal imaging technology, OCT-AFI, will be used to image sites on the cervix, the endocervical canal and vulva. The imaging probe is small enough, it can be inserted into the endocervical canal for imaging. The probe can also be placed in a conformable holder that can be shaped to conform the the folds of the vulva for vulvar imaging. The resultant images will be compared to histology images.

The objectives are to determine

1. feasibility of the technology in imaging vulva and its capability in detecting vulvar intraepithelial neoplasias
2. feasibility in imaging cervix from endocervical canal to transformation zone to ectocervix
3. if combined OCT with AFI increases the sensitivity of detecting high grade lesions in the cervix compared to just AFI alone (previous work was AFI alone).

DETAILED DESCRIPTION:
The multimodal optical imaging technology, OCT-AFI, has demonstrated the ability to image the small peripheral airways of the lung, allowing for high resolution of structural and functional details of airway tissue and the vasculature. Through the OCT (optical coherence tomography) component, the bronchial epithelium can be visualized and its thickness quantifiable. Micro invasion of the basement membrane can be seen in the acquired images. The AFI (autofluorescence imaging) component showed the vascular network, areas of pulmonary fibrosis and areas with loss of endogenous fluorescence beside pulmonary nodules.

The investigators anticipate OCT-AFI to be able to see subsurface structures in the cervix and vulva as well. Through previous work, the investigators found AFI to be sensitive to detecting high grade cervical lesions but the technology was confounded by normal subsurface tissue structures. By combining OCT with AFI, the investigators anticipate a higher sensitivity to detecting high grade lesions on the cervix than with just AFI. The OCT-AFI imaging probe is also small enough to fit into the endocervical canal and will allow for imaging of neoplasias that originate in the canal. These abnormalities are on the rise. Vulvar neoplasias are also on the rise and visually difficult to identify and determine surgical margins. OCT-AFI may help clinicians locate and determine the extent of vulvar lesions.

The objectives are to determine

1. feasibility of the technology in imaging vulva and its capability in detecting carcinoma and vulvar intraepithelial neoplasias
2. feasibility in imaging complete cervix from endocervical canal to transformation zone to ectocervix
3. if combined OCT with AFI increases the sensitivity of detecting high grade lesions in the cervix compared to just AFI alone (previous work was AFI alone).

This study will image 10 subjects for endocervical canal and ectocervix sites. Another 10 subjects will be imaged for vulvar sites. Imaging will not affect where standard of care biopsies will be taken from. Imaging results will be correlated with histology.

No statistical analysis will be performed. This feasibility study will look at the quality and utility of the acquired image sets. If possible, the investigators will quantify the images in terms of epithelium thickness, basement membrane location, presence of vasculature and sub-epithelial structures.

ELIGIBILITY:
Inclusion Criteria:

* indicates understanding of study
* provides informed consent to participate
* 18 years or older
* not pregnant and have negative urine pregnancy test
* be scheduled for initial visit colposcopy for cervix or vulva or LEEP (loop electrosurgical excision procedure) for treatment of abnormalities on cervix at the Women's Clinic at Vancouver General Hospital (VGH)

Exclusion Criteria:

* breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from VGH Women's Clinic. They will have a scheduled appointment for an initial visit colposcopy for cervix or vulva (that is, a biopsy will be done) or they will have a scheduled LEEP appointment.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Determine ease of use of OCT-AFI in imaging cervix or vulva lesions. | Total imaging session of cervix and canal or vulva should take no more than 5 minutes
  The ability to image complete cervix including endocervical canal or vulvar lesions in one continuous imaging run will indicate the device is feasible for use in the clinical setting for cervix and vulva. Note whether a complete image scan was collected or not after each imaging session.

SECONDARY OUTCOMES:
Correlate OCT-AFI images with histology images | 6 months
  Correlate sub-epithelial structures seen in OCT-AFI with histology images
Quantify OCT-AFI images by examining epithelial thickness | 6 months
  Measure epithelial thickness along entire scanned image. Units of measure in millimeters.
Locate basement membrane invasion and loss of normal endogenous fluorescence | 6 months
  Locate basement membrane in OCT-AFI images and note presence or absence of invasion. Note presence or absence of fluorescence in epithelial layer in images.
Note extent of vasculature and its features | 6 months
  Make notes regarding vasculature patterns seen in the OCT-AFI images.

CONTACTS AND LOCATIONS:
Overall Officials: Calum MacAulay, Ph.D., Principal Investigator — British Columbia Cancer Agency
Locations (1):
- Vancouver General Hospital Women's Clinic, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee AM, Ohtani K, Macaulay C, McWilliams A, Shaipanich T, Yang VX, Lam S, Lane P. In vivo lung microvasculature visualized in three dimensions using fiber-optic color Doppler optical coherence tomography. J Biomed Opt. 2013 May;18(5):50501. doi: 10.1117/1.JBO.18.5.050501. PMID 23625308
- [Background] Pahlevaninezhad H, Lee AM, Ritchie A, Shaipanich T, Zhang W, Ionescu DN, Hohert G, MacAulay C, Lam S, Lane P. Endoscopic Doppler optical coherence tomography and autofluorescence imaging of peripheral pulmonary nodules and vasculature. Biomed Opt Express. 2015 Sep 30;6(10):4191-9. doi: 10.1364/BOE.6.004191. eCollection 2015 Oct 1. PMID 26504665
- [Background] Pahlevaninezhad H, Lee AM, Shaipanich T, Raizada R, Cahill L, Hohert G, Yang VX, Lam S, MacAulay C, Lane P. A high-efficiency fiber-based imaging system for co-registered autofluorescence and optical coherence tomography. Biomed Opt Express. 2014 Aug 6;5(9):2978-87. doi: 10.1364/BOE.5.002978. eCollection 2014 Sep 1. PMID 25401011